CLINICAL TRIAL: NCT07046520
Title: Effects of High-Intensity Interval Training on Plasma Volume, Muscle Damage, and Aerobic Performance in Overweight Adolescent Females
Brief Title: Effects of HIIT on Plasma Volume and Aerobic Capacity in Obese Adolescent Girls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: High Institute of Sports and Physical Education of Kef (Other)
Responsible Party: Principal Investigator, Wissal Abassi, Principal Investigator, High Institute of Sports and Physical Education of Kef
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HIIT-ADO-2025-TN
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2024-12

CONDITIONS: Hematologic Test
Keywords: Obesity; High-Intensity Interval Training; Adolescent Girls; Creatine Kinase; Plasma Volume Variation; Aerobic Capacity; Erythrocytes
MeSH Terms: conditions — Obesity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity interval training group (Experimental): High-intensity interval training group performed four series of 15-second runs at 90-105% of the maximal aerobic speed (MAS) interspersed with 15 seconds of active recovery at 5O% MAS.
  Interventions: Behavioral: High intensity interval training
- Control group (No Intervention): No training intervention was intended for the control group.

INTERVENTIONS:
Behavioral: High intensity interval training — HIIT protocol was performed three times per week over a 10-week period, totaling 30 sessions. HIIT sessions included: (1) a standardized warm-up of five minutes of continuous jogging at 50%MAS, followed by five minutes of dynamic mobility and activation drills such as high-knee skips, high-knee running, and butt kicks. (2) a HIIT training session, consisted of four series of 15-second runs at 90-105% of the maximal aerobic speed (MAS) interspersed with 15 seconds of active recovery and (3) a cool-down of five minutes of static stretching.
  Arms: High-intensity interval training group

SUMMARY:
The goal of this clinical trial is to investigate the impact of high-intensity interval training (HIIT) program on body composition, hematological parameters, plasma volume variations (PVV), muscle damage markers, and aerobic capacity in overweight/obese adolescent girls. The main question it aims to answer is: Does HIIT reduce risk factors associated obesity diseases by modulating body composition and hematological parameters and increasing PVV? Researchers will compare HIIT (designed to the experimental group) to nontraining intervention (designed to the control group) to see if the training program works to enhance physiological health and reduce risk factors associated with obesity in this population. Participants in the experimental (HIIT group) group will: underwent HIIT at 90-105% maximal aerobic speed (MAS), three times a week.

Participants in control group will : not perform any physical training and maintain their usual daily activities.

DETAILED DESCRIPTION:
Obesity during adolescence is linked to adverse changes in body composition, aerobic fitness, and blood health. High-intensity interval training (HIIT) is a promising strategy to improve these outcomes. However, its effects on hematological markers, plasma volume, and muscle damage in overweight/obese adolescent girls remain unclear. This study aimed to investigate the effects of HIIT on body composition, hematological parameters, plasma volume variations (PVV), muscle damage markers, and aerobic capacity in this population.Twenty-eight overweight/obese girls (16.21±0.92) were randomly assigned to a HIIT group (n=14) or control group (n=14). The 10-week HIIT protocol consisted of 4×6×15s running at 90-105% maximal aerobic speed (MAS) with 15s of active recovery at 50% MAS (3 sessions/week). Pre/post assessments included body composition, hematological markers, muscle damage markers, and aerobic fitness. Plasma volume was estimated post-intervention in both group.

ELIGIBILITY:
Inclusion Criteria:

* Females.
* Aged between 15 and 17 years.
* BMI greater than or equal to the 95th percentile for their age.

Exclusion Criteria:

* Pharmacological treatments or medical conditions that could interact with the protocol (e.g.,hypertension, diabetes, cardiac, orthopedic, neuromuscular, or neurological disorders).
* Hormone replacement therapy or therapies for obesity.
* Irregular menstrual cycle.
* Restrictive diet or use of dietary supplements or engagement in any structured physical training either currently or during the previous three months.
* Withdrawal of consent.
* Non-compliance with study procedures.
* Insufficient data for analysis.

Ages: 15 Years to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Female
Enrollment: 28 (Actual)
Dates: Start 2024-12-09 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Erythrocytes | At baseline and at week 11 (end of intervention period).
  Blood levels of erythrocytes were collected from a blood sample (5 ml) and analyzed using a multichannel automated hematology analyzer (XN450; Sysmex, Norderstedt, Germany).
Hemoglobin | At baseline and at week 11 (end of intervention period).
  Blood levels of hemoglobin were collected from a blood sample (5 ml) and analyzed using a multichannel automated hematology analyzer (XN450; Sysmex, Norderstedt, Germany).
Hematocrit | At baseline and at week 11 (end of intervention period).
  Blood levels of hematocrit were collected from a blood sample (5 ml) and analyzed using a multichannel automated hematology analyzer (XN450; Sysmex, Norderstedt, Germany).
Mean corpuscular volume | At baseline and at week 11 (end of intervention period).
  Blood levels of mean corpuscular volume were collected from a blood sample (5 ml) and analyzed using a multichannel automated hematology analyzer (XN450; Sysmex, Norderstedt, Germany).
Mean corpuscular hemoglobin content | At baseline and at week 11 (end of intervention period).
  Blood levels of mean corpuscular hemoglobin content were collected from a blood sample (5 ml) and analyzed using a multichannel automated hematology analyzer (XN450; Sysmex, Norderstedt, Germany).
Mean hemoglobin concentration | At baseline and at week 11 (end of intervention period)
  Blood levels of mean hemoglobin concentration were collected from a blood sample (5 ml) and analyzed using a multichannel automated hematology analyzer (XN450; Sysmex, Norderstedt, Germany).
Creatine kinase | At baseline and at week 11 (end of intervention period).
  Serum concentrations of creatine kinase are measured from a blood sample (5 ml) using a Beckman Coulter AU480 Chemistry Analyzer (France).
Lactate dehydrogenase | At baseline and at week 11 (end of intervention period).
  Serum concentrations of lactate dehydrogenase are measured from a blood sample (5 ml) using a Beckman Coulter AU480 Chemistry Analyzer (France).
Plasma volume variations | Plasma volume variations (PVV) was calculated at week 11 (end of intervention period) under two conditions (High intensity interval training and No training intervention [control group] ).
  Plasma volume variations (PVV) was calculated based on measured hematocrit (Ht) and hemoglobin (Hb) values according to the method developed by Costill and Fink (1974). %PVV=100 ×[(HbA/HbB) ×(100 - HtB) / (100 - HtA)] - 1, where 0 is the value measured before training program and 1 is the value measured after training program.
Body weight | At baseline and at week 11 (end of intervention period).
  Body weight (kg) was recorded , with barefoot and lightly dressed subjects, using an electronic scale (Tanita BC-533, Tokyo, Japan).
Height | At baseline
  Height (m) was determined using a standard stadiometer (Holtain Ltd., UK).
Body fat | At baseline and at week 11 (end of intervention period)
  Body fat (%) was recorded using an electronic scale (Tanita BC-533, Tokyo, Japan).
Body mass index | At baseline and at week 11 (end of intervention period).
  Body mass index (kg/m²) was calculated as weight (kg) divided by height squared (m²).
Waist circumference | At baseline and at week 11 (end of intervention period).
  Waist circumference (cm) was measured to the nearest 0.1 cm using a non-deformable anthropometric tape, placed horizontally at the midpoint between the inferior margin of the last palpable rib and the superior border of the iliac crest, with the participant standing upright and breathing normally.
Maximal aerobic speed | At baseline and at week 11 (end of intervention period).
  Maximal aerobic speed was determined using the Vameval test (Cazorla,1990).
Maximal oxygen consumption (VO2max) | At baseline and at week 11 (end of intervention period).
  Maximal oxygen consumption (VO2max) were determined using the Vameval test (Cazorla,1990).
Maximal heart rate (HRmax) | At baseline and at week 11 (end of intervention period).
  Maximal heart rate maximum (HRmax) was recorded at the final stage of the Vameval test (Cazorla,1990) using a Polar heart rate monitor (Polar S810, Kempele, Finland).

CONTACTS AND LOCATIONS:
Overall Officials: Wissal abassi, Dr, Principal Investigator — Research Unit "Sport Sciences, Health and Movement"(UR22JS01) High Institute of Sport and Physical Education of Kef, University of Jendouba, 7100 Kef, Tunisia.
Locations (1):
- High Institute of Sports and Physical Education of Kef, El Kef, Boulifa, Tunisia

IPD SHARING:
Plan to Share IPD: No
For confidentiality reasons, all data from this study are available upon request.